CLINICAL TRIAL: NCT04404153
Title: Non-Invasive Home Neurostimulation for Mild to Moderate Alzheimer's Disease: Double-Blind, Sham Controlled Randomized Clinical Trial
Brief Title: Neurostimulation for Cognitive Enhancement in Alzheimer's Disease
Acronym: NICE-AD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: MJHS Institute for Innovation in Palliative Care (Other); Stony Brook University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-11274; R01AG068167 (NIH)
Record Dates: First submitted 2020-05-22; First posted 2020-05-27 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Alzheimer's Disease; transcranial direct current stimulation (tDCS)
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Active tDCS (Experimental): The active tDCS will involve 30-minutes of direct current at intensity of 2 milliamperes (mA).
  Interventions: Device: tDCS device model Soterix mini-CT (Soterix Medical Inc., New York, NY) programed to deliver active tDCS.
- Sham tDCS (Sham Comparator): Sham stimulation consists of the direct current ramped up to 2mA over 30 seconds, ramped down over 30 seconds and stay at 0 current for the remaining application period.
  Interventions: Device: tDCS device model Soterix mini-CT (Soterix Medical Inc., New York, NY) programed to deliver sham tDCS.

INTERVENTIONS:
Device: tDCS device model Soterix mini-CT (Soterix Medical Inc., New York, NY) programed to deliver active tDCS. — At-home remotely supervised tDCS delivered over the dorsolateral prefrontal cortex with the anode on the left, cathode on the right, at an intensity of 2 mA, delivered for 30 minutes five times per week (Monday-Friday) for 26 weeks (6 months).
  Arms: Active tDCS
Device: tDCS device model Soterix mini-CT (Soterix Medical Inc., New York, NY) programed to deliver sham tDCS. — Sham treatment will consist of the current ramped up to 2mA over 30 seconds, ramped down over 30 seconds and stay at 0 current for the remaining time of the 30-minute application period five times per week (Monday-Friday) for 26 weeks (6 months).
  Arms: Sham tDCS

SUMMARY:
The prevalence of Alzheimer's Disease (AD) is rising, but existing medications provide only modest control of cognitive decline and associated symptoms, and novel therapies are urgently needed. This randomized sham-controlled trial will determine if an innovative low-risk remotely-supervised transcranial Direct Current Stimulation (tDCS) applied over the area of the dorsolateral prefrontal cortex for 30 minutes at the intensity of 2 mA five times per week for 6 months at home can improve cognitive performance and symptoms and modulate neuroimaging markers of neuroplasticity in 100 patients with mild to moderate AD. If effective, this novel intervention can substantially enhance AD symptom management at home, improve quality of life of AD patients and their families, and reduce burden associated with this debilitating illness.

DETAILED DESCRIPTION:
The hallmark of Alzheimer's Disease (AD) is cognitive decline with varied associated symptoms and signs. Unfortunately, there is no cure as yet for AD. Available treatments, including 5 FDA-approved medications, have limited efficacy in terms of slowing pathological progression or controlling the symptoms and signs of cognitive decline in AD patients. Given the high burdens and costs of AD, and the therapeutic limitations, the development of novel treatment approaches for AD is of the highest importance for patients, families, medical providers, and society. This randomized controlled trial will determine if innovative, low-risk neurostimulation at home for 6 months can improve cognitive performance and symptoms in patients with mild to moderate AD.

The primary objective is to determine the effects produced by 6 months of active tDCS or sham delivered over dorsolateral prefrontal cortex (DLPFC) in home settings on global cognitive performance (assessed by ADAS-Cog test - primary outcome), and secondarily on executive control/spatial selective attention (Eriksen Flanker Test), depressed mood (Geriatric depression scale), quality of life (Quality of Life Questionnaire-Alzheimer's Disease), and patient satisfaction with both the device and procedure (Neurostimulation User's Survey), in mild-to-moderate AD patients (n=100). The investigators also aim to determine functional and structural brain connectivity/network changes in response to the study intervention using functional Magnetic Resonance Imaging (fMRI; during rest and during executive function tasks), diffusion-weighted imaging (DWI), and multivariate covariance-based analytic approaches. Lastly, the investigators aim to examine time characteristics (durability) of the tDCS behavioral and neuroplasticity effects for up to 3 months following the intervention period.

The intervention will consist of remotely supervised active tDCS stimulation and sham tDCS stimulation over the area of the dorsolateral prefrontal cortex, applied at home for 30 minutes 5 times per week for 6 months. Participants randomized to the active tDCS will receive at each application 30 minutes of direct current stimulation at the intensity of 2 mA. Participants randomized to the sham group will receive sham tDCS which consists of current ramped up to 2mA over 30 seconds, ramped down over 30 seconds and stay at 0 current for the remaining time of the 30-minute application.

ELIGIBILITY:
Inclusion Criteria:

1. Community-dwelling male or female of age 60 and older.
2. AD diagnosed by neurologists or geriatricians at our dementia and geriatric clinical sites. Clinicians will review the medical records of all potential cases to ensure the patients meet established clinical criteria for AD, and also examine individuals as needed to further establish the diagnosis. Mild-to moderate stage AD as determined by study clinicians using the Clinical Dementia Rating Scale (CDR). The CDR is a 5-point scale used to characterize six domains of cognitive and functional performance applicable to AD: Memory, Orientation, Judgment & Problem Solving, Community Affairs, Home & Hobbies, and Personal Care. The necessary information to make each rating is obtained through a semi-structured interview of the patient and a reliable informant (e.g., family member). A CDR score of 0.5 or 1 is rated as mild severity and a score of 2 is rated as moderate severity. The investigators selected mild to moderate AD patients as our target population as they are the most prevalent AD severity group referred to our clinics, increasing generalizability. This mild to moderate AD group is also most likely to be cared for in the community and at home, in contrast to more advanced or severe AD stages, which are more prevalent in institutional settings (and will be the focus of our future studies).
3. If on dementia medication regimen, the regimen is stable for at least 4 weeks prior to enrollment. The investigators will not restrict clinicians from starting, adjusting or stopping dementia medications over the intervention period in keeping with the pragmatic nature of our trial, but will account for medications in both groups in our analysis.
4. Able to speak and understand English or Spanish at a level sufficient undergo the study procedures and testing protocols.
5. Willing to complete an MRI (exclusions relevant to neuroimaging are described below).
6. Able to provide Informed Consent (or able to provide assent with a legal surrogate providing informed consent.)

Exclusion Criteria:

1. Unstable medical or major psychiatric illnesses or unstable treatments for medical or major psychiatric illnesses. Any medical or psychiatric diagnosis is permitted as long as it has been clinically stable for at least 3 months, reflected in part by stability of treatments for at least 3 months, and is expected on the basis of clinical judgment to be in a stable phase that will likely extend for 6 months.
2. History of head trauma, seizures, brain surgery, stroke or cancer affecting head, metal implants in the head or neck, compromised integrity or sensitivity of the skin at or near locations where electrodes will be placed (e.g., eczema, severe rashes, blisters, open wounds, burn including sunburns, cuts or irritation).
3. Currently participating in another intervention study or using neurostimulation device.
4. Exclusions specific to neuroimaging procedure: the presence of any surgically implanted metallic devices, such as aneurysm clips or pacemakers that would be a safety contraindication for MRI. Subjects with large amounts of dental or surgical hardware in the head and neck will be excluded because magnetic susceptibility effects will lead to severe image artifacts in these subjects' images. Due to the confined space of the MRI magnet, subjects with a known history of claustrophobia will also be excluded as will subjects with weight >350lbs or waist circumference >55 inches.
5. Must not be currently receiving or have received (or completed) within the past 3 months any monoclonal antibody treatment for Alzheimer's

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Global Cognitive Performance | Baseline, at 6 months (immediately after the 6-month intervention)
  Change in The Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-Cog) was developed as an outcome measure for dementia interventions; its primary purpose was to be an index of global cognition in response to therapies. It assesses multiple cognitive domains across 11 items: Word Recall Task, Naming Objects and Fingers, Following Commands, Constructional Praxis, Ideational Praxis, Orientation, Word Recognition Task, Remembering Test Directions, Spoken Language, Comprehension and Word-Finding Difficulty. The score ranges from 0 to 70. A 4-point ADAS-cog change at 6 months is clinically meaningful.

SECONDARY OUTCOMES:
Multiple-Domain Cognitive Dysfunction | Baseline, at 6 months (immediately after the 6-month intervention), at 7 months (1 month post-intervention) and 9-months (3 months post-intervention).
  The Digit Symbol Substitution Test (a subtest of the Wechsler Adult Intelligence Scale - Revised) is a measure of attention, transcription and speed of processing. Scoring is based on the total number of correct responses generated during a 90-sec time interval. Higher values reflect better outcome.
Executive control/spatial selective attention | Baseline, at 6 months (immediately after the 6-month intervention), at 7 months (1 month post-intervention) and 9-months (3 months post-intervention).
  The Flanker Test is a measure of speed of processing, attention and inhibitory control. Scoring is based on accuracy and reaction time. Lower values reflect better outcome.
Quality of Life Scale | Baseline, at 6 months (immediately after the 6-month intervention), at 7 months (1 month post-intervention) and 9-months (3 months post-intervention).
  The Quality of Life - Alzheimer's Disease, self-reported includes 13 items representing physical, social and psychological well-being. The administration takes about 5 minutes.
Depressive Symptoms | Baseline, at 6 months (immediately after the 6-month intervention), at 7 months (1 month post-intervention) and 9-months (3 months post-intervention).
  Changes in depressive symptoms assessed using the 15 item Geriatric Depression Scale, scores range from 0 (not depressed) to 15 (depressed).
Tolerability of the study intervention: number of side effects and adverse events | Baseline, at 6 months (immediately after the 6-month intervention), at 7 months (1 month post-intervention) and 9-months (3 months post-intervention).
  Determined as number of side effects and adverse events related, probably related or possibly related to the study intervention.
Patient's satisfaction: 8-item tDCS User Survey | Baseline, at 6 months (immediately after the 6-month intervention)
  Patient's satisfaction with the study intervention determined from the 8-item tDCS User Survey at the end of the intervention. Each item of the Survey is a brief statement and a respondent indicates if s/he Strongly Agree, Agree, Neither Agree or Disagree, Disagree or Strongly Disagree with the statement. Higher number of Agree/Strongly Agree ratings reflects higher satisfaction with the tDCS procedure.
Functional Neuroplasticity-Digit Symbol Substitution | Baseline, at 6 months (immediately after the 6-month intervention) and 9-months (3 months post-intervention).
  The investigators will examine intervention-related changes in functional activation/deactivation networks during Digit Symbol Substitution Test. The investigators predict tDCS-related changes in functional/deactivation relative to sham - particularly in dorsolateral prefrontal cortex and associated networks.
Functional Neuroplasticity - Flanker Interference Task | Baseline, at 6 months (immediately after the 6-month intervention) and 9-months (3 months post-intervention).
  The investigators will examine intervention-related changes in functional activation/deactivation networks during Flanker tests. The investigators predict tDCS-related changes in functional/deactivation relative to sham - particularly in dorsolateral prefrontal cortex and associated networks.

OTHER OUTCOMES:
Structural Neuroplasticity | Baseline, at 6 months (immediately after the 6-month intervention) and 9-months (3 months post-intervention).
  The investigators propose to explore pre-post changes in structural connectivity as a function of tDCS. Structural changes in white matter integrity have been observed following tDCS in another study. Based on these initial findings, the investigators propose to monitor structural changes in white matter integrity (fractional anisotropy) using FreeSurfer's v.6.0 Tracts Constrained by Underlying Anatomy (TRACULA).
Durability of Global Cognitive Performance | Baseline and 9-months (3 months post-intervention).
  Change in The Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-Cog) was developed as an outcome measure for dementia interventions; its primary purpose was to be an index of global cognition in response to therapies. It assesses multiple cognitive domains across 11 items: Word Recall Task, Naming Objects and Fingers, Following Commands, Constructional Praxis, Ideational Praxis, Orientation, Word Recognition Task, Remembering Test Directions, Spoken Language, Comprehension and Word-Finding Difficulty. The score ranges from 0 to 70. A 4-point ADAS-cog change at 6 months is clinically meaningful.

CONTACTS AND LOCATIONS:
Overall Officials: Joe Verghese, MD, Principal Investigator — Stony Brook University; Lara Dhingra, PhD, Principal Investigator — Metropolitan Jewish Health System; Mirnova Ceide, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gulley E, Verghese J, Blumen HM, Ayers E, Wang C, Portenoy RK, Zwerling JL, Weiss E, Knotkova H. Neurostimulation for cognitive enhancement in Alzheimer's disease (the NICE-AD study): a randomized clinical trial. Neurodegener Dis Manag. 2021 Aug;11(4):277-288. doi: 10.2217/nmt-2020-0061. Epub 2021 Jul 9. PMID 34240627

DOCUMENTS (1):
  • Informed Consent Form (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/53/NCT04404153/ICF_000.pdf